CLINICAL TRIAL: NCT00874783
Title: Derivation of Induced Pluripotent Stem Cells from Somatic Cells Donated by Patients with Neurological Diseases for the Study of the Pathogenesis of the Disorders and Development of Novel Therapies
Brief Title: Development of IPS from Donated Somatic Cells of Patients with Neurological Diseases
Status: Recruiting | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: 0599-08-HMO-CTIL
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Neurodegenerative Disorders
Keywords: Amyotrophic Lateral Sclerosis; Familial Dysautonomia; Parkinson's Disease; Alzheimer's Disease; Age Related Macular Degeneration; Retinitis Pigmentosa; Huntington's Disease; Machado - Joseph Disease; SMA - Spinal Muscular Atrophy; Ataxia Telangiectasia
MeSH Terms: conditions — Neurodegenerative Diseases; Amyotrophic Lateral Sclerosis; Dysautonomia, Familial; Parkinson Disease; Alzheimer Disease; Macular Degeneration; Retinitis Pigmentosa; Huntington Disease; Muscular Disorders, Atrophic; Muscular Atrophy, Spinal; Ataxia Telangiectasia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — donation of a skin specimen of up to 10mm in diameter from skin which will be removed in a surgical operation from a patient who is scheduled to undergo an operation for medical reasons and with no relation to the study at hand.
Oversight: Data Monitoring Committee: No

SUMMARY:
Human fibroblasts and possibly other human somatic cells may be reprogrammed into induced pluripotent stem (iPS) cells by the forced expression of transcription factors (1-5). The iPS cells seem to share many properties with human embryonic stem cells.

Induced pluripotent stem cells potentially may be useful in the future as an unlimited source of cells for transplantation.

The major goal of the project is to develop human iPS cells from cell cultures from skin biopsies or the patient's hair. The iPS cells will be developed primarily for modeling diseases and drug discovery as well as basic research, and for developing the technology that may eventually allow the use of iPS cells for future transplantation therapy. The iPS cells developed in the course of this application are not intended for use in transplantation therapy. Future development of iPS cells for clinical transplantation therapies will be subjected to the appropriate authorization by ethical and regulatory committees.

DETAILED DESCRIPTION:
The derivation of human iPS cells (1-5) open new avenues to model human diseases since it may now be possible to develop iPS cells from the fibroblasts or other somatic cells of patients with various conditions. These iPS cells may be directed to differentiate into the cells which are affected in specific conditions. Abnormalities in the development of the affected cells as well as altered survival or function of the cells may be studied. Thus iPS cells may serve as an invaluable model for the study of the pathogenesis of human diseases and may also serve for the development of new drugs, and high throughput screening of molecules for toxic or therapeutic effects.

In addition to the great potential of iPS cells for disease modelling and transplantation therapy, the cells may have broad applications in basic research in various areas such as reprogramming, basic development and others.

At present, it is still unclear whether the properties of iPS cells are identical to those of hESCs. Initial data suggest that human iPS cells are indeed similar to hESCs in their phenotype, epigenetic status of pluripotent self-specific genes, telomerase activity, gene expression profile and in their capability to differentiate into progeny of the three germ layers both in vitro and in vivo in teratomas (2, 3, 5). In the mouse system, directed differentiation of iPS cells into bone marrow repopulating hematopoietic stem cells and functional dopaminergic neurons was demonstrated (6, 7). However, incomplete silencing of the constitutive expression of the transcription factors that were used to induce reprogramming can probably interfere with differentiation (1). Further studies are required to confirm that the developmental potential and biological properties of iPS cells are identical to hESC.

Currently, retroviral vectors are most commonly used to introduce and express the transgenes which reprogram the somatic nucleus (1-5). The use of retroviral vectors, which integrate into the host cell genome, may cause hazardous insertion mutagenesis. Moreover, the use of potentially oncogenic transcription factors, such as c-Myc, significantly limits the clinical use of human iPS cells for future cell therapy. However, successful derivation of iPS cells was demonstrated without the forced expression of c-Myc. The decreased efficiency of reprogramming, in the absence of overexpressed c-Myc, may be improved by molecules which act via epigenetic mechanisms. Moreover, successful derivation of iPS cells was recently reported with the use of non-integrating adeno viral vectors or repeated transfections. Thus it appears that with further developments, it may be possible in the future to safely induce pluripotent cells from somatic cells for therapeutic applications.

ELIGIBILITY:
Inclusion Criteria:

* Donors suffering from different (specified) neurodegenerative disorders scheduled to undergo surgery for medical reasons or will donate a single or a few hairs--to be removed intact from the scull or other areas in the body.
* Healthy donors scheduled to undergo surgery for medical reasons or will donate a single or a few hairs--to be removed intact from the scull or other areas in the body.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 120 donors to cover 10 different neurodegenerative disorders (previously specified) based on 10 donors per disorder and 20 healthy control donors.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2009-04 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin E Reubinoff, MD, PhD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Ein Kerem, Jerusalem, Israel, Israel

REFERENCES:
- [Background] Yu J, Vodyanik MA, Smuga-Otto K, Antosiewicz-Bourget J, Frane JL, Tian S, Nie J, Jonsdottir GA, Ruotti V, Stewart R, Slukvin II, Thomson JA. Induced pluripotent stem cell lines derived from human somatic cells. Science. 2007 Dec 21;318(5858):1917-20. doi: 10.1126/science.1151526. Epub 2007 Nov 20. PMID 18029452